CLINICAL TRIAL: NCT06795048
Title: A Phase IIIb/IV, Multicenter, Randomized, Open-Label, Two-Arm Study to Investigate the Efficacy, Safety, and Durability of Faricimab Administered up to Every 24 Weeks in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: A Study to Determine the Efficacy, Safety, and Durability of Faricimab in Participants With Neovascular Age-Related Macular Degeneration
Acronym: CONSTANCE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MR45638; 2024-517545-13-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-01-24; First posted 2025-01-27 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Neovascular Age-related Macular Degeneration (nAMD)
MeSH Terms: interventions — faricimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Faricimab Early Treat & Extend Regimen (Experimental)
  Interventions: Drug: Faricimab
- Arm B: Faricimab Modified Treat & Extend Regimen (Experimental)
  Interventions: Drug: Faricimab

INTERVENTIONS:
Drug: Faricimab — Participants will receive 6-mg faricimab intravitreal (IVT) injections in the study eye according to the dosing regimen for the study arm to which they are randomized.
  Other Names: RO6867461; VABYSMO®

SUMMARY:
This study is a Phase IIIb/IV, multicenter, randomized, two-arm, open-label 100-week study to investigate the efficacy, safety, and durability of intravitreal 6-mg faricimab administered at up to 24-week intervals in patients with neovascular age-related macular degeneration (nAMD) that are treatment-naïve in the study eye.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy as determined by medical evaluation that includes medical history and physical examination
* Agreement to adhere to the contraception requirements described in the protocol

Ocular Inclusion Criteria for Study Eye:

* Active treatment-naïve macular neovascularization (MNV) secondary to age-related macular degeneration (AMD), confirmed by the investigator based on the presence of intraretinal fluid (IRF) or subretinal fluid (SRF) affecting the central subfield on optical coherence tomography (OCT)
* BCVA of 83 to 24 letters, inclusive (20/25 to 20/320 approximate Snellen equivalent, using the early treatment diabetic retinopathy study [ETDRS] protocol and addressed at the initial testing distance of 4 meters on Day 1)
* Sufficiently clear ocular media and adequate pupillary dilation to allow acquisition of good quality retinal images to confirm diagnosis

Exclusion Criteria:

Ocular Exclusion Criteria for Study Eye:

* MNV due to causes other than nAMD, such as ocular histoplasmosis, trauma, pathological myopia, angioid streaks, choroidal rupture, or uveitis
* Retinal pigment epithelial tear involving the macula on Day 1
* Current vitreous hemorrhage on Day 1
* Prior periocular pharmacological or IVT treatment (including faricimab, anti-vascular endothelial growth factor [VEGF], or complement inhibitor medication) for other retinal diseases

Ocular Exclusion Criteria for Fellow (Non-Study) Eye:

* Participants who have a nonfunctioning fellow (non-study) eye, defined as either BCVA of hand motion or worse, or no physical presence of non-study eye (i.e., monocular), at both the screening and study Day 1 visits

Ocular Exclusion for Both Eyes:

* History of idiopathic or autoimmune associated uveitis in either eye
* Active ocular inflammation or suspected or active ocular or periocular infection in either eye on study Day 1

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2027-09-16 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Best-Corrected Visual Acuity (BCVA) Score Averaged Over Weeks 44, 48, and 52 | Baseline and average of Weeks 44, 48, and 52

SECONDARY OUTCOMES:
Change from Baseline in BCVA Score Averaged Over Weeks 92, 96, and 100 | Baseline and average of Weeks 92, 96, and 100
Change from Baseline in BCVA Score Over Time | From Baseline to Week 100
Percentage of Participants Avoiding a Loss of ≥15 Letters in BCVA from Baseline Over Time | From Baseline to Week 100
Percentage of Participants with BCVA Snellen Equivalent of 20/40 or Better Over Time | From Baseline to Week 100
Percentage of Participants with BCVA Snellen Equivalent of 20/200 or Worse Over Time | From Baseline to Week 100
Change from Baseline in Central Subfield Thickness (CST) Averaged Over Weeks 44, 48, and 52 | Baseline and average of Weeks 44, 48, and 52
Change from Baseline in CST Averaged Over Weeks 92, 96, and 100 | Baseline and average of Weeks 92, 96, and 100
Change from Baseline in CST Over Time | From Baseline to Week 100
Percentage of Participants on Different Treatment Intervals at Weeks 52 and 100 | Weeks 52 and 100
Incidence and Severity of Ocular Adverse Events | From first study treatment to Week 100
Incidence and Severity of Non-Ocular Adverse Events | From first study treatment to Week 100

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (67):
- United States (11):
  - Orange County Retina Medical Group, Santa Ana, California
  - Florida Retina Institute, Orlando, Florida
  - Ctr for Retina & Macular Dis, Winter Haven, Florida
  - Retinal Vitreal Consultants, Chicago, Illinois
  - University Retina and Macula Associates, PC, Lemont, Illinois
  - New England Retina Consultants, Springfield, Massachusetts
  - Sierra Eye Associates, Sparks, Nevada
  - Retina Associates of New Jersey, Teaneck, New Jersey
  - Vision Research Center at Eye Associates of New Mexico, Albuquerque, New Mexico
  - Charles Retina Institute, Germantown, Tennessee
  - Retina Consultants of Texas, Schertz, Texas
- Australia (6):
  - Strathfield Retina Clinic, Strathfield, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - Adelaide Eye and Retina Centre, Adelaide, South Australia
  - Centre For Eye Research Australia, East Melbourne, Victoria
  - Retina Specialists Victoria, Rowville, Victoria
  - The Lions Eye Institute, Nedlands, Western Australia
- Canada (5):
  - St. Joseph's Health Care, London, Ontario
  - Retina Institute of Ottawa, Ottawa, Ontario
  - Toronto Retina Institute, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Hopital du Saint Sacrement, Québec, Quebec
- China (6):
  - Peking University People's Hospital, Beijing
  - West China Hospital of Sichuan University, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou
  - Eye and ENT hospital, Fudan University, Shanghai
  - Tongji Hosp, Tongji Med. Col, Huazhong Univ. of Sci. & Tech, Wuhan
- France (6):
  - Centre Retine Gallien, Bordeaux
  - Hopital Edouard Herriot - CHU Lyon, Lyon
  - Centre Ophtalmologique de L'Odeon, Paris
  - Hopital Lariboisiere, Paris
  - Centres Ophtalmologique St Exupéry, Saint-Cyr-sur-Loire
  - Clinique de l'Union, Saint-Jean
- Germany (5):
  - Augenzentrum Prof. Koch GmbH, Frankfurt
  - Medizinische Hochschule Hannover, Klinik für Augenheilkunde, Hanover
  - Augenzentrum am St Franziskus-Hospital, Münster
  - Universitatsklinikum Ulm, Augenklinik und Poliklinik, Ulm
  - Universitätsklinikum Würzburg, Augenklinik und Poliklinik, Würzburg
- Italy (6):
  - Azienda ospedaliero universitaria Policlinico Riuniti di Foggia;SC Oculistica, Foggia, Apulia
  - Azienda ospedaliero - universitaria Sant'Andrea;UOC Oculistica, Rome, Lazio
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Ospedale San Giuseppe, Milan, Lombardy
  - Azienda Ospedaliera Universitaria "Luigi Vanvitelli";UOC Oculistica, Napoli, Sicily
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Torrette - Ancona, The Marches
- Singapore (2):
  - Singapore Eye Research Institute, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (6):
  - Pusan National University Hospital, Busan
  - Yeungnam Univ. Hospital, Daegu
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (5):
  - Hospital General de Catalunya, Sant Cugat de Valles, Barcelona
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Oftalvist, Burjassot, Valencia(España), Valencia
  - Clinica Baviera, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Zhongzheng Dist.
- United Kingdom (6):
  - Cardiff and Vale University Health Board, Cardiff
  - St James University Hospital, Leeds
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - NewcastleUniversity& The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing